CLINICAL TRIAL: NCT07345169
Title: Studies on the Immunological and Inflammatory Determinants Associated With the Prognosis of Patients Admitted to Intensive Care
Brief Title: IMMUNOREA - Immunological and Inflammatory Determinants Associated With the Prognosis of Intensive Care Patients
Acronym: IMMUNOREA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM U942 (Unknown); Société Française d'Anesthésie et de Réanimation (Other); French Society for Intensive Care (Other); European Society of Intensive Care Medicine (Other); ZOLL Foundation, Fondation Les Gueules Cassées (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP250001; 2025-A00002-47 (Other: IDRCB)
Record Dates: First submitted 2025-09-05; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Intensive Care Patients; Critical Illness Requiring Intensive Care - Sepsis; Critical Illness Requiring Intensive Care - Acute Brain Injury; Critical Illness Requiring Intensive Care - Major Surgery; Critical Illness Requiring Intensive Care - Polytrauma
Keywords: Sepsis; Critical illness; Intensive care; Immunology; Inflammation; Transcriptomics; scRNAseq; Flow cytometry; Nosocomial infections; Prognosis
MeSH Terms: conditions — Critical Illness; Sepsis; Inflammation; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational physiopathological study aimed at evaluating the immunological and inflammatory determinants associated with the prognosis of patients admitted to intensive care units (ICU). The study will establish multidimensional models predicting one-year survival and the occurrence of nosocomial infections.

Patients admitted to ICU undergo routine biological sampling. In addition to these, minimal supplementary samples will be collected for immunological and inflammatory biomarker analysis at admission, day 1, day 4, day 8, ICU discharge or day 28, and at 12 months. Additional samples may be taken during clinically significant events (nosocomial infections, complications).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to ICU within 24 hours

Exclusion Criteria:

* Moribund patient (ECOG=4)
* Legal protection (guardianship/curatorship)
* Uninsured patients
* Pre-existing immunosuppression (active/recent cancer, hematologic disease, autoimmune disease, organ transplant, HIV)
* Pregnant or breastfeeding women
* Participation in another interventional trial
* Patients under AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥ 18 years old) admitted to intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival of patients admitted to intensive care. | 12 months
  Difference in overall survival between ISU patients with different immunological and inflammatory profiles upon completion of the 12-month follow-up period.
Multidimensional flow cytometry leukocyte profiling | Change from baseline to 12 months
  The isolated cell samples will be analyzed to determine the absolute number and percentage of B cells, monocytes, CD4+ and CD8+ T cells, CD3+CD56+ NKT cells, and NK cells
Inflammatory profile of ICU patients | Change from baseline to 12 months
  Inflammation-related protein biomarkers will be analyzed using Olink assay

SECONDARY OUTCOMES:
Change in SOFA Score | Change from baseline to day 7
  Sequential Organ Failure Assessment (SOFA) Score included the degree of dysfunction of six organ systems (Respiratory, Cardiovascular, Liver, Renal, Coagulation, Neurologic). Minimum score = 0 maximum score = 24. Higher scores indicate greater degree of dysfunction.
Transcriptomic (scRNAseq) profiling of isolated leukocytes | Change from baseline to12 months
  Change in the transcriptome of leukocytes isolated from blood, bronchoalveolar lavage fluid (BAL), cerebrospinal fluid (CSF), urine, and tissues, as measured by single cell RNA-sequencing using Flex technology

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP Laribosière Hospital, Anesthesia and Critical Care Departement, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available upon reasonable request, after publication of primary results, for research purposes only.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code